CLINICAL TRIAL: NCT04236531
Title: Source-monitoring Processes and Risk for Psychosis
Brief Title: Source-monitoring & Psychosis
Acronym: SOURIPSY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-A02499-48
Record Dates: First submitted 2020-01-06; First posted 2020-01-22 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Psychosis
Keywords: source-monitoring; at-risk; MRI; neuroimaging
MeSH Terms: conditions — Psychotic Disorders | interventions — Neuropsychological Tests; Neuroimaging

STUDY DESIGN:
Intervention Model Description: Three groups of participants will be recruited: individuals at ultra-high risk for psychosis, first-episode psychosis patients and healthy controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- individuals at ultra-high risk for psychosis (UHR) (Experimental): 30 individuals meeting the UHR criteria according to the "Comprehensive Assessment of at-risk mental state" (CAARMS) will be recruited and will complete cognitive task and MRI scan
  Interventions: Other: Cognitive tests and neuroimaging
- patients with first episode psychosis (FEP) (Experimental): 30 patients with first episode psychosis (FEP) will be recruited and will complete cognitive task and MRI scan
  Interventions: Other: Cognitive tests and neuroimaging
- healthy controls (Sham Comparator): 30 healthy individuals will be recruited and will complete cognitive task and MRI scan
  Interventions: Other: Cognitive tests and neuroimaging

INTERVENTIONS:
Other: Cognitive tests and neuroimaging — comparison of cognitive performances and brain anatomy

SUMMARY:
Source-monitoring is a cognitive process that refers to the ability to remember the source of an information. Some studies have showed source-monitoring deficits in patients with schizophrenia as well as in individuals at ultra-high risk for psychosis (UHR) and in first-episode psychosis patients (FEP). Source-monitoring deficits have thus been proposed as a potential early risk factor for psychosis. However, further studies are needed to better characterize this deficit.

The aim of this project is to investigate source-monitoring performances in UHR, FEP patients and healthy controls (HC) and to characterize these deficits in terms of brain anatomy, basic auditory processes and social functioning.

DETAILED DESCRIPTION:
Ninety participants will be included in the study: 30 UHR, 30 FEP and 30 healthy controls. All the participants will complete a standardized source-monitoring task, an MRI acquisition (3D-T1 anatomical scan), a tone-matching task as well as a socio-demographic and clinical evaluation including an assessment of the social functioning.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women aged between 18 and 30
* Having given their written informed consent
* French speakers and readers
* Absence of hearing impairments (or tinnitus) that could prevent the successful completion of tasks involving listening to sounds or words
* Absence of visual impairments that could prevent the successful completion of tasks involving reading on the screen
* For the healthy control group, no history of previous diagnosed psychiatric disorders (according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders - DSM5), absence of relatives diagnosed with spectrum disorder schizophrenia and bipolar disorder (DSM5), absence of psychotic prodromes measured by a score of less than 6 in the "prodromal questionnaire" - PQ-16 (Ising et al., 2012), absence of drug treatments (except oral contraception).
* For the UHR group, meeting the UHR criteria according to the "Comprehensive Assessment of at-risk mental state" (CAARMS).
* For the FEP group, presenting with daily psychotic symptoms for at least a week.

Exclusion Criteria:

* Do not consent to be included in the study
* Contraindication to MRI scan
* History of neurological disease
* Pregnancy
* Being under tutorship or curatorship
* Having developed musical abilities (that is, regularly practicing a musical instrument)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Source-monitoring performances | one day
  Scores obtained at a source-monitoring task (Brunelin et al., 2006)

SECONDARY OUTCOMES:
Confidence in source-monitoring judgements | one day
  Confidence in source-monitoring judgements will be measured using a visual analogue scale (0-100)
Grey matter volume | one day
  Grey matter volume will be assessed with a structural MRI scan (3D-T1) followed by morphometry analyses.
Brain gyrification | one day
  Brain gyrification will be assessed with a structural MRI scan (3D-T1) followed by gyrification analyses.
Basic auditory performances | one day
  scores at the Tone Matching Task (Strous et al., 1995)
Working memory performances | one day
  scores at a working memory task (Barrouillet et al., 2004)
Social functioning | one day
  score at the "personal and social performance scale" (0-100)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier le Vinatier, Bron, France

IPD SHARING:
Plan to Share IPD: Undecided